CLINICAL TRIAL: NCT01050660
Title: Low Dose Parenteral Fat for Prevention of Parenteral Nutrition Associated Cholestasis in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of California, Los Angeles (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Richard Ehrenkranz, Professor of Pediatrics, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIC# 0902004803
Record Dates: First submitted 2009-12-23; First posted 2010-01-15 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Parenteral Nutrition-Associated Liver Disease
Keywords: Parenteral nutrition associated liver disease; Direct bilirubin; Intravenous fat emulsion; Very low birth weight infants; PNAC
MeSH Terms: interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 gm/kg/day intravenous lipid emulsion (Active Comparator)
  Interventions: Other: Intravenous fat emulsion
- Intravenous Fat Emulsion-restricted (Experimental)
  Interventions: Other: Restriction of intravenous fat emulsion to 1 gm/kg/d

INTERVENTIONS:
Other: Intravenous fat emulsion — An infusion of intravenous fat will start at 0.5 grams/kg on the first day of life, with increments of 0.5 -1.0 grams/kg every day, until a total dose of 3 grams/kg is reached.
  Arms: 3 gm/kg/day intravenous lipid emulsion
Other: Restriction of intravenous fat emulsion to 1 gm/kg/d — Intravenous fat will be started at 0.5 grams/kg on the first day of life and then increase to a dose of 1gram/kg/day the next day. There will be no further increase in the amount of intravenous fat.
  Arms: Intravenous Fat Emulsion-restricted

SUMMARY:
The goal of the study is to determine if parenteral nutrition-associated cholestasis (PNAC) is related to the amount of parenteral (intravenous) fat administered to premature babies until full enteral nutrition is achieved.

DETAILED DESCRIPTION:
In the neonatal intensive care unit, parenteral nutrition is widely used to provide protein, energy, vitamins and minerals to infants who cannot accept enteral feeds.

Intravenous fat emulsion is an important component of parenteral nutrition because of the important caloric supply that it brings, but also for the essential fatty acids (linoleic and linolenic acid) that it provides. Because intravenous fat emulsion is the only supply of essential fatty acids, at least until the enteral feeds are established, there is a minimum of fat that has to be administered with at least 0.25g/kg /day for preterm babies and 0.1g/kg/day for term infants (Lee EJ, 1993). The maximal dose of intravenous fat safe to administer is difficult to determine. Although in larger preterm infants intravenous fat is tolerated well based on measurement of serum triglycerides, there are still question regarding tolerance in extremely low birth weight infants.

Parenteral nutrition has been associated with the development of liver disease-parenteral nutrition associated liver disease (PNALD). PNALD can range from cholestasis and a transient elevation of liver enzymes to more severe forms including fibrosis, liver cirrhosis and hepatic failure. Cholestasis, defined as hyperbilirubinemia with a direct bilirubin above 2 mg/dL or more than 15% of total bilirubin, is a hepatocellular injury of the liver that manifests after the administration of parenteral nutrition for at least two weeks. The mechanism by which the liver injury occurs is unknown and probably multifactorial. Risk factors associated with the development of PNAC include: prematurity, low birth weight, absence of enteral feeds, bacterial sepsis, necrotizing enterocolitis, prolonged use of parenteral nutrition, and multiple surgical procedures on the gastro-intestinal tract. In addition, many of the nutrients contained in parenteral nutrition, have been linked with the development of cholestasis.

Specific factors associated with intravenous fat emulsions that have been related to PNAC include : phytosterols, the rate of administration of the intravenous emulsion, the total amount of fat administered and toxic metabolites of intravenous fat emulsions.

The total amount of lipids was found to be a risk factor for cholestasis in children on long-term parenteral nutrition and decreased amount of fat was recommended for the prevention of this hepatic complication (Colomb V, 2000). In the adult population parenteral lipid intake of less than 1gr/kg of body weight decreased the risk of cholestasis in parenteral nutrition treated patients (Cavicchi, 2000).

Current Nutritional Management for VLBW infants in the NBSCU:

The administration of parenteral nutrition to all the preterm babies with a gestational age less than or equal to 29 weeks' is standard practice in the NBSCU for infants not receiving full enteral nutrition. Fat, as an integral part of the intravenous alimentation, is started in the first day of life at a dose of 0.5 grams/kg/day of an 20% fat emulsion(eg, Lyposyn II, Abbott Laboratories Chicago, IL). The amount of fat is then gradually increased by 0.5-1 grams/kg/day to total amount of 3 grams/kg/day as tolerated. The tolerance is checked by measuring serum triglyceride level the morning after 3 grams/kg/day has been reached for the first time serum triglyceride level ≤200 mg/dl are accepted for infants ≤52 weeks postmenstrual age. If the serum triglyceride level is >200 mg/dL, the intravenous fat emulsion is reduced for 24 hours, then the triglyceride level is checked again to ensure that it has dropped below 200 mg/dL. The fat emulsion is then restarted at 1-1.5 grams/kg/day and the serum triglyceride level is monitored as it is slowly increased.

Enteral nutrition is started initially as minimal enteral feedings, also called non-nutritive feedings, usually by 48±12 hours of age with about 12 ml/kg/day. The feedings are then advanced as tolerated with the goal to reach full enteral nutrition (>120 ml/kg/day) between 14-21days of life. As the enteral volumes reach 1/3, 1/2, and 2/3 of the total daily fluid volume, the rate of administration of the lipid emulsion is decreased in steps (ie, from 2 grams/kg/day to 1.5 to 1.0) , until the intravenous fat emulsion is stopped.

As part of standard NBSCU management guidelines screening of liver function consists of measuring serum direct bilirubin level after the baby has been on TPN for 10 days to two weeks and then biweekly, if PN continues. In addition, if the direct bilirubin level is greater than 2.5mg/dL, then liver enzymes will be checked .

Study Procedure:

All preterm babies with a gestational age less than or equal to 29 weeks' born at YNHH who will receive intravenous fat emulsion as part of their nutrition management are eligible to participate in the study. The parents of these babies will be approached during the first 24 hours of life, regarding the possible participation in the study. After informed consent will be obtained, the subjects will be randomized by YNHH Investigator pharmacy to one of the two groups: intervention (restricted intravenous fat intake) and control (standard intravenous fat intake).

Therefore, the purpose of this study will be to determine if PNAC is related to the amount of parenteral fat administered to premature babies until full enteral nutrition is reached.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than or equal to 29 weeks' gestation
* Age less than 48 hours

Exclusion Criteria:

* Congenital intrauterine infection, known to be associated with liver involvement and cholestasis
* Known structural liver abnormalities that are associated with cholestasis
* Known genetic disorders: trisomy 21, trisomy 13 and trisomy 18
* Inborn errors of metabolism
* Infants meeting the criteria for terminal illness (eg, pH < 6.8 > 2 hours)
* Inability to obtain informed consent

Ages: 12 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2009-06; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Ehrenkranz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Lee EJ, Simmer K, Gibson RA. Essential fatty acid deficiency in parenterally fed preterm infants. J Paediatr Child Health. 1993 Feb;29(1):51-5. doi: 10.1111/j.1440-1754.1993.tb00440.x. PMID 8461181
- [Background] Colomb V, Jobert-Giraud A, Lacaille F, Goulet O, Fournet JC, Ricour C. Role of lipid emulsions in cholestasis associated with long-term parenteral nutrition in children. JPEN J Parenter Enteral Nutr. 2000 Nov-Dec;24(6):345-50. doi: 10.1177/0148607100024006345. PMID 11071594
- [Background] Boyd GW. An investigation of the prolonged pressor response to renin in the nephrectomized rat. Clin Sci Mol Med Suppl. 1976 Dec;3:151s-153s. doi: 10.1042/cs051151s. PMID 1071594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bewtween May 2009 -November 2012- infants born and admitted to NICU were enrolled.
Groups:
- 3 gm/kg/Day Intravenous Lipid Emulsion: Intravenous fat emulsion : An infusion of intravenous fat will start at 0.5 grams/kg on the first day of life, with increments of 0.5 -1.0 grams/kg every day, until a total dose of 3 grams/kg is reached.
- Intravenous Fat Emulsion-restricted: Restriction of intravenous fat emulsion to 1 gm/kg/d : Intravenous fat will be started at 0.5 grams/kg on the first day of life and then increase to a dose of 1gram/kg/day the next day. There will be no further increase in the amount of intravenous fat.
Period: Overall Study
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Started | 67 | 69
Completed | 67 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 67 | 69 | 136
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 41 | 46 | 87
Region of Enrollment [Number; unit: participants]
  United States | 67 | 69 | 136
Gestational age at enrollement [Mean (Standard Deviation); unit: weeks] — Gestational age, in full completed weeks at enrollement.
  weeks | 26.4 (1.8) | 26.6 (1.8) | 26.5 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: The Presence of Cholestasis at Age of 28 Days or When Full Enteral Nutrition is Achieved, Whichever is Longer.
Time Frame: 28 days of age or when full enteral nutrition is acheived, whichever is longer
Population: Incidence of PNALD at Yale and UCLA NICU prior to the start of the study was around 40%.
  Our goal was to decrease incidence by 50%/ Alpha of 5%/ Power of 80% We calculated a sample size of 65 infants in each group
Measure: Number; unit: participants who developed Cholestasis
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
participants who developed Cholestasis | 39 | 45

2. Secondary Outcome: Mortality Rate- Death Rate Before Discharge From the Hospital
Time Frame: Discharge from the Newborn ICU
Measure: Number; unit: participants
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
participants | 5 | 6

3. Secondary Outcome: Incidence of Bronchopulmonary Dysplasia (BPD)
Time Frame: 36 weeks PMA or discharge home,whichever comes first
Measure: Number; unit: participants who developed BPD
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
participants who developed BPD | 27 | 26

4. Secondary Outcome: Incidence of Necrotizing Enterocolitis (NEC)
Time Frame: At discharge from Newborn ICU
Measure: Number; unit: participants who developed NEC
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
participants who developed NEC | 8 | 11

5. Secondary Outcome: Incidence of Retinopathy of Prematurity (ROP)
Time Frame: At discharge from Newborn ICU
Measure: Number; unit: participants who developed ROP
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
participants who developed ROP | 7 | 9

6. Secondary Outcome: Late Onset Sepsis
Description: Bloodstream infection, defined as a positive blood culture obtained after 72 hours of life.
Time Frame: At the discharge from Newborn ICU
Measure: Number; unit: participants who developed LOS
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
participants who developed LOS | 3 | 5

7. Secondary Outcome: Length of Stay
Description: Defines time to discharge or death.
Time Frame: At discharge from Newborn ICU/death
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
Days | 81.5 [64.3 to 108.8] | 87 [66.5 to 110.8]

8. Secondary Outcome: Anthropometric Measurements(Body Weight)
Description: Change in body weight measurement reported in g/week
Time Frame: At age of 28 days and at discharge
Measure: Mean (Standard Deviation); unit: g/week
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
g/week | 66.6 (34) | 62.9 (39)

9. Secondary Outcome: Anthropometric Measurements(Length)
Description: Change in body length measurement reported in cm/week
Time Frame: At age of 28 days and at discharge
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
cm/week | 0.8 (0.5) | 0.9 (0.5)

10. Secondary Outcome: Anthropometric Measurements(Head Circumference)
Description: Change in head circumference measurement reported in cm/week
Time Frame: At age of 28 days and at discharge
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Number analyzed (Participants) | 67 | 69
cm/week | 0.5 (0.3) | 0.6 (0.3)

ADVERSE EVENTS:
Arm/Group | 3 gm/kg/Day Intravenous Lipid Emulsion | Intravenous Fat Emulsion-restricted
Serious Adverse Events (participants affected / at risk) | 5/67 | 6/69
Other Adverse Events (participants affected / at risk) | 0/67 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 gm/kg/Day Intravenous Lipid Emulsion (N=67) | Intravenous Fat Emulsion-restricted (N=69)
Mortality prior to discharge (General disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No